CLINICAL TRIAL: NCT00587275
Title: A Double-Blind, Randomized, Placebo-Controlled Crossover Study to Assess the Efficacy of AST-120 in Patients With Gastroesophageal Reflux Disease (GERD) Who Continue to be Symptomatic on a Standard Dose of Proton Pump Inhibitor (PPI)
Brief Title: Safety and Efficacy of AST-120 in Patients With GERD Who Continue to be Symptomatic on a Standard Dose of PPI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for lack of enrollment
Sponsor: Ocera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AST013
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — AST 120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AST-120, 2 gram sachets
  Interventions: Drug: AST-120
- 2 (Placebo Comparator): Celphere CP-305, stained to match appearance of AST-120 in 2g sachets.
  Interventions: Drug: Celphere CP-305

INTERVENTIONS:
Drug: AST-120 — Oral, sachet, 2 grams daily for 4 weeks
  Arms: 1
Drug: Celphere CP-305 — Oral, sachet, 2 grams daily for 4 weeks
  Arms: 2

SUMMARY:
The purpose of this project is to test how safe and how well AST-120, an investigational product, works in treating too much acid in the stomach. Patients will be randomly assigned to one of two groups, AST-120 or a placebo for the first four weeks of the study. The patients will be switched to the other group (AST-120 or placebo)for the following four weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, crossover trial where 20 patients with confirmed persistent GERD symptoms (at least twice weekly) after a standard course of PPI, with abnormal bile reflux levels but normal esophageal acid exposure are randomized to initially receive either AST-120 or placebo for a period of 4 weeks after a two week screening period. After a washout period of one week, patients will cross over to the opposite blinded treatment.

The experimental drug AST-120 is composed of black, odorless spherical carbon particles in 2g sachets (aluminum foil pouches). The placebo consists of microcrystalline cellulose spheres, Celphere CP-305, stained to match the appearance of AST-120, in 2g sachets (aluminum foil pouches). Both AST-120 and placebo are oral (taken by mouth) preparations. Both are tasteless. Take the product, patients will tear open the sachet, drop the contents directly on their tongue and wash it down with 8 ounces of water.

Patients will continue to receive the previously prescribed PPI throughout the duration of the trial. In addition, patients will be allowed up to 6 Gelusil tablets daily as a "rescue medication".

Patients will be expected to participate in approximately 5 in-clinic visits. During these visits, patients will undergo a number of tests including: comprehensive physical, hematology panel, a urine pregnancy test for pre-menopausal females, completion of the Gastroesophageal Reflux Disease Symptom Assessment Scale (GSAS) and Short-Form-36 (SF-36)Quality of Life Form and an upper endoscopy will be performed to determine the extent of esophageal inflammation.

Patients will be allowed to continue on their previously prescribed PPI with no changes and may take up to 6 Gelusil tablets per day. The following therapies must be discontinued and should not be taken during the trial: H2receptor antagonists, NSAIDs, Baclofen and Antacids (OTC or prescription).

ELIGIBILITY:
Inclusion Criteria:

* Body weight 40 to 136 kg (88 to 300 lbs)
* Recent history of GERD related symptoms (at least twice weekly) confirmed during screening.
* Recent history of 8 week PPI treatment without significant improvement
* Abnormal bilirubin level as assessed by Bilitec
* Normal esophageal pH value (pH<4.0 for <4.2% of the time calculated over a 24 hour period)
* Platelet count (thrombocytes) >100,000/µL
* Normal Hgb and Hct levels
* Able and willing to comply with all protocol procedures for the planned duration of the study
* Able and willing to understand, sign and date an informed consent document, and authorize access to protected health information.
* Females must be postmenopausal, surgically incapable of bearing children, or practicing a reliable method of birth control (hormonal contraceptives, intrauterine devices, spermicide and barrier). Partner/spouse sterility may also qualify at the Investigator's discretion. Females of child-bearing potential must have a negative urine pregnancy test at baseline.

Exclusion Criteria:

* Concurrent GI or other pathology which could interfere with the course of the study (e.g., erosive esophagitis, malabsorption, cirrhosis, ascites, bleeding ulcer, diabetes, scleroderma, non-GI myopathy or neuropathy etc.) Note: patients with Barrett's esophagus (short segment defined as < 3 cm) can be included.
* Patients with cancer or undergoing chemotherapy for the treatment of cancer
* Patients with a history of upper GI surgery
* Patients with GERD complications such as stricture of the esophagus
* Contraindication to continued PPI treatment
* Patients requiring the concomitant use of NSAIDs for the duration of the study
* Uncontrolled systemic disease
* Diagnosis of a psychiatric disorder within the past 2 years and not on a stable dose of medications for at least 6 months
* Other major physical or psychiatric illness in previous 6 months as determined by the treating physician
* Known hypersensitivity or contraindication to any component of the test product (study drug) or diagnostics used
* Participation in another study within eight (8) weeks prior to randomization
* Unable to attend all visits required by the protocol
* Pregnant, breast feeding, or planning to become pregnant during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Reduction in the severity of GERD symptoms in patients receiving AST-120 assessed by comparing the symptom scores on the GSAS. | 8 weeks
Safety endpoint is adverse events (AEs)deemed possibly, probably, or definitely related to treatment with investigational product. | 8 weeks

SECONDARY OUTCOMES:
Reduction in severity of GERD symptoms in patients receiving AST-120 assessed by patient self assessment using a daily diary. | 8 weeks
Percent days without heartburn. | 8 weeks
Percent daytime period without heartburn. | 8 weeks
Percent change in SF-36 score. | 8 weeks
Esophageal bilirubin levels as measured by Bilitec. | 8 weeks
Amount of rescue medication (Gelusil) taken per day. | 8 weeks
Changes in clinical laboratory tests from baseline. | 8 weeks
Prior and concomitant medications. | 8 weeks
Physical examination, vital signs (blood pressure, heart rate, respiration rate and temperature). | 8 weeks
GI tolerability (diarrhea, constipation, etc). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — Southern Arizona VA Health Care System
Locations (1):
- Southern Arizona VA Health Care System and University of Arizona Health Sciences Center, Tucson, Arizona, United States

REFERENCES:
- [Background] Xu XR, Li ZS, Zou DW, Xu GM, Ye P, Sun ZX, Wang Q, Zeng YJ. Role of duodenogastroesophageal reflux in the pathogenesis of esophageal mucosal injury and gastroesophageal reflux symptoms. Can J Gastroenterol. 2006 Feb;20(2):91-4. doi: 10.1155/2006/498142. PMID 16482234
- [Background] Fennerty MB. Review article: alternative approaches to the long-term management of GERD. Aliment Pharmacol Ther. 2005 Dec;22 Suppl 3:39-44. doi: 10.1111/j.1365-2036.2005.02711.x. PMID 16303036
- [Background] Fass R, Shapiro M, Dekel R, Sewell J. Systematic review: proton-pump inhibitor failure in gastro-oesophageal reflux disease--where next? Aliment Pharmacol Ther. 2005 Jul 15;22(2):79-94. doi: 10.1111/j.1365-2036.2005.02531.x. PMID 16011666
- [Background] Fukuda Y, Takazoe M, Sugita A, et al. The treatment with an oral spherical adsorptive carbon (AST-120) improves anal fistula, PDAI and CDAI scores - A randomized double-blind placebo controlled trial. Abstract #765 presented at Digestive Disease Week meeting, Los Angeles, CA May 24, 2006
- [Background] Yamazaki Z, Fujimori T, Yoshimoto T, et al. Effect of Oral Adsorbent on Animal Models of Hepatic Failure 92(2):331-335, 1980
- [Background] Araki Y, Tsujikawa T, Andoh A, Sasaki M, Fujiyama Y, Bamba T. Therapeutic effects of an oral adsorbent on acute dextran sulphate sodium-induced colitis and its recovery phase in rats, especially effects of elimination of bile acids in gut lumen. Dig Liver Dis. 2000 Nov;32(8):691-8. doi: 10.1016/s1590-8658(00)80332-1. PMID 11142579